CLINICAL TRIAL: NCT06463002
Title: Ambulatory Blood Pressure Control and Cognition in Patients With Obstructive Sleep Apnea
Brief Title: Ambulatory Blood Pressure Control and Cognition in Patients With Obstructive Sleep Apnea (AMPLE)
Acronym: AMPLE
Status: Not yet recruiting | Type: Observational
Sponsor: National University Hospital, Singapore (Other)
Collaborators: Alexandra Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2023/01017
Record Dates: First submitted 2024-06-12; First posted 2024-06-17 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive Sleep Apnea; Hypertension; Cognitive impairment
MeSH Terms: conditions — Sleep Apnea, Obstructive; Hypertension; Cognitive Dysfunction | interventions — Blood Pressure Monitoring, Ambulatory

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- OSA treated: Patients with OSA treated with CPAP for at least six months
  Interventions: Diagnostic Test: Ambulatory blood pressure monitoring and Montreal Cognitive Assessment
- OSA untreated: Patients with OSA not treated with CPAP
  Interventions: Diagnostic Test: Ambulatory blood pressure monitoring and Montreal Cognitive Assessment
- non-OSA: Patients underwent a sleep study and were diagnosed not to have OSA
  Interventions: Diagnostic Test: Ambulatory blood pressure monitoring and Montreal Cognitive Assessment

INTERVENTIONS:
Diagnostic Test: Ambulatory blood pressure monitoring and Montreal Cognitive Assessment — Noninvasive tests to assess blood pressure control and cognition

SUMMARY:
To compare the blood pressure control and cognitive responses of three groups of patients: those diagnosed with Obstructive Sleep Apnea (OSA) and treated with Continuous Positive Airway Pressure (CPAP) for at least six months, those diagnosed with OSA but not treated, and those without OSA.

DETAILED DESCRIPTION:
This study is designed as an observational, cross-sectional investigation at the National University Hospital and Alexandra Hospital. The research aims to enroll 50 eligible patients in each of the three groups (OSA treated, OSA untreated, and non-OSA, totaling 150 participants). The recruited participants will undergo ambulatory blood pressure monitoring (ABPM) and the Montreal Cognitive Assessment (MoCA). ABPM is a widely used, noninvasive method to determine patients' blood pressure control. MoCA is a widely used screening tool designed to assess cognitive function and detect mild cognitive impairment or early signs of dementia. The MoCA evaluates various cognitive domains, including attention, memory, language, visuospatial abilities, executive functions, and orientation. It consists of a series of tasks and questions that assess different aspects of cognitive functioning, such as drawing specific shapes, recalling words or numbers, and performing simple calculations. A trained healthcare professional will administer the digital version of the MoCA, which usually takes less than 30 minutes to complete. The MoCA has been validated for use in diverse populations and has shown good sensitivity in detecting mild cognitive impairment. The maximum score on the MoCA is 30. Lower scores may indicate potential cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* Known OSA (AHI >/=15 events/ hour, based on sleep study) on CPAP treatment for at least six months (n=50)
* Known OSA (AHI >/=15 events/ hour, based on sleep study) NOT on CPAP treatment (n=50)
* Known non-OSA (AHI <15 events/ hour, based on sleep study) (n=50)

Exclusion Criteria:

* Known-OSA on non-CPAP treatment (e.g., mandibular advancement device, surgery, or hypoglossal nerve stimulation),
* Heart failure,
* Atrial fibrillation, or acute coronary syndrome in the prior 3 months
* Dementia (based on the medical record)
* Previous stroke
* Non-English-speaking subjects
* Pregnant and lactating women

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals who fulfil the inclusion criteria but not the exclusion criteria will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
24-hour mean systolic blood pressure | Within 4 weeks after consent (one time)
  A 24-hour ambulatory blood pressure monitoring will be performed
Montreal Cognitive Assessment (MoCA) | Within 4 weeks after consent (one time)
  Montreal Cognitive Assessment scale (0-30). Lower the scale means more severe cognitive impairment

SECONDARY OUTCOMES:
Office systolic blood pressure | Within 4 weeks after consent (one time)
  Office blood pressure will be record
Epworth Sleepiness Scale | Within 4 weeks after consent (one time)
  Epworth Sleepiness Scale (4-24). Higher scale means more severe daytime sleepiness
Nocturnal blood pressure dipping | Within 4 weeks after consent (one time)
  Percentage of Participants with >10% drop in nocturnal systolic blood pressure based on the ambulatory BP monitoring
24-hour systolic blood pressure <130 mmHg | Within 4 weeks after consent (one time)
  24-hour systolic blood pressure <130 mmHg based on the ambulatory BP monitoring
24-hour systolic blood pressure <120 mmHg | Within 4 weeks after consent (one time)
  24-hour systolic blood pressure <120 mmHg based on the ambulatory BP monitoring
Montreal Cognitive Assessment (MoCA) <27 | Within 4 weeks after consent (one time)
  Prevalence of participants with Montreal Cognitive Assessment (MoCA) <27
Montreal Cognitive Assessment (MoCA) <20 | Within 4 weeks after consent (one time)
  Prevalence of participants with Montreal Cognitive Assessment (MoCA) <20
MoCA score <27 (for those with >10 years of education) and <26 (for those with ≤10 years of education) | Within 4 weeks after consent (one time)
  Prevalence of participants with MoCA score <27 (for those with >10 years of education) and <26 (for those with ≤10 years of education)

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital, Singapore, SG, Singapore

IPD SHARING:
Plan to Share IPD: Yes
Plan to make individual participant data (IPD) available to other researchers at least 5 years after study completion, subjected to final approval by the PI
Supporting Information: CSR
Time Frame: At least 5 years after study completion
Access Criteria: Plan to make individual participant data (IPD) available to other researchers at least 5 years after study completion, subjected to final approval by the PI